CLINICAL TRIAL: NCT07026006
Title: Effects of Active Release Versus Strain-Counter-strain Technique on Pain, Range of Motion, Cranio-vertebral Angle, and Disability in Patients With Non-Specific Neck Pain
Brief Title: Active Release Versus Strain-Counter-strain Technique in Patients With Non-Specific Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Junad- REC/RCR&AHS 24/0141
Record Dates: First submitted 2025-06-11; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Neck Pain
Keywords: Neck Pain; Soft Tissue Therapy; Trigger points; Cervicalgia; Posterior Cervical Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group A (Experimental): Active Release Technique
  Interventions: Other: Active Release Technique
- Treatment Group B (Active Comparator): Strain-counterstrain
  Interventions: Other: Strain-counterstrain

INTERVENTIONS:
Other: Active Release Technique — Patients will receive Active Release Technique (ART) protocol will be applied to 4 muscles Including; trapezius, levator scapulae, sternocleidomastoid (SCM), and suboccipital muscles (for 15 minutes)
  Arms: Treatment Group A
Other: Strain-counterstrain — Patients will receive Strain-counterstrain (SCS) protocol will be applied to 4 muscles Including the trapezius, levator scapulae, sternocleidomastoid (SCM), and suboccipital muscles for 15 minutes.
  Arms: Treatment Group B

SUMMARY:
The study design will be a randomized clinical trial (RCT) aims to compare the effects of Active Release Technique and Strain-Counterstrain on pain, range of motion, cranio-vertebral angle, and disability in patients with non-specific neck pain. Data will be collected from Safi Teaching Hospital, Faisalabad, Pakistan. Using a non-probability purposive sampling method, participants aged 18-45 years with localized cervical pain and stiffness will be selected based on inclusion and exclusion criteria. The inclusion and exclusion criteria will be; Participants aged 18-45, both male and female, experiencing neck pain for at least 2 months, with palpable taut bands in upper trapezius and SCM, active trigger points in upper trapezius, levator scapulae, and SCM, NPRS score >3/10 for neck region, and localized pain/stiffness in cervical spine (C3-C7) without upper limb radiculopathy, confirmed by negative Spurling's test, upper limb tension test, and shoulder abduction test. Subjects will be excluded if presented with a history of Participants who received myofascial treatment in the preceding month or have a diagnosis of fibromyalgia, KNGF Clinical Practice Guideline Grade III or IV, or neurological deficits.

Participants will be equally divided into 2 groups using a random number generator table. Group A will receive Active Release Technique, while Group B will receive Strain-Counterstrain. Both groups will also receive hot packs, superficial neck muscles stretching, and neck isometrics. Outcome measures, including the Numerical Pain Rating Scale for pain, goniometer for range of motion, cranio-vertebral angle measurement, Neck Disability Index, will be assessed at baseline and after four weeks. Ethical approval will be obtained from the Ethical Committee of Riphah International University, and informed consent will be secured from all participants. The outcomes will focus on pain intensity, cervical range of motion, cranio-vertebral angle, and disability, Data analysis will be performed using SPSS version 25. The findings are expected to provide valuable insights into the comparative efficacy of these manual therapy techniques, informing clinical practice and improving patient outcomes in the management of non-specific neck pain.

DETAILED DESCRIPTION:
Neck discomfort is defined as pain that is felt anywhere along the posterior cervical spine, which runs from the superior nuchal line to the first thoracic spinous process. (According to IASP).The annual prevalence of neck pain varies widely over the world, from 30% to 50%. This can significantly impair the quality of life and disable individuals who are impacted.With the potential to significantly affect people, their families, communities, and healthcare systems, neck discomfort is regarded as the fourth most common disability in the world.

Neck pain is a prevalent musculoskeletal disorder affecting a significant portion of the global population at some point in their lives. It is estimated that up to 70% of people will experience neck pain during their lifetime. According to the global burden of disease in the Mediterranean region, the point prevalence of neck pain was estimated as 34.31 per 1000 in Pakistan.

Neck pain is often classified into specific and non-specific categories. Non-specific neck pain lacks a definitive cause and is frequently associated with poor posture, muscle strain, or minor injuries. It can become chronic, leading to prolonged discomfort and disability. Chronic neck pain affects daily activities, work performance, and overall well-being, making effective management essential.

In Pakistan, the prevalence of non-specific neck pain mirrors global trends, affecting a considerable portion of the population. Studies indicate that around 34% of the population in Pakistan experiences non-specific neck pain, driven by factors such as sedentary lifestyles, poor posture, and ergonomic issues in workplaces.

The rationale for this study is grounded in the high prevalence and significant impact of neck pain on individuals' quality of life and overall well-being. Non-specific neck pain affects a considerable portion of the population, leading to chronic pain and disability. Current treatments, while effective, often vary in their outcomes, necessitating a comparison of different therapeutic techniques. This study focuses on comparing the effects of Active Release Technique and Strain-Counterstrain, two promising manual therapy approaches. To figure out their efficacy in reducing pain, improving range of motion, and enhancing postural alignment. By investigating these methods, this study seeks to provide novel insights into their comparative effectiveness, which has been underexplored.

The findings will inform clinical practice, potentially leading to more personalized and effective treatment plans. Additionally, the study aims to address the socioeconomic burden of neck pain by improving patient outcomes and reducing healthcare costs. Through rigorous methodology and comprehensive analysis, this research aspires to contribute significantly to the field of manual physical therapy and enhance the management of non-specific neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years
* Both male and female
* Patients with neck pain for at least 2 months
* Palpable taut bands in upper trapezius, SCM
* ATrPs in upper trapezius, levator scapulae, SCM
* NPRS score is >3/10 on NPRS for neck region
* Individuals with a Craniovertebral angle less than 53
* Individuals having grade 2 severity of neck pain according to KNGF Guidelines
* Localized pain/stiffness in cervical spine (C3-C7) without upper limb radiculopathy
* Diagnostic Tests: Negative Spurling's test, upper limb tension test, and shoulder abduction test

Exclusion Criteria:

* Myofascial treatment in the preceding month
* Diagnosis of fibromyalgia
* Congenital problems
* Trigger point injections
* Individuals with KNGF Clinical Practice Guideline Grade III and IV severity of neck pain
* Respiratory disease and joint disease
* Neurological deficit

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-28 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain rating Scale | Baseline, 4th Week
Neck Disability Index | Baseline, 4th Week
Craniovertebral Angle | Baseline, 4th Week
Cervical Range of Motion | Baseline, 4th Week

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil ur Rehman, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Campos TF, Maher CG, Steffens D, Fuller JT, Hancock MJ. Exercise programs may be effective in preventing a new episode of neck pain: a systematic review and meta-analysis. J Physiother. 2018 Jul;64(3):159-165. doi: 10.1016/j.jphys.2018.05.003. Epub 2018 Jun 19. PMID 29908853
- [Background] Cabrera-Martos I, Rodriguez-Torres J, Lopez-Lopez L, Prados-Roman E, Granados-Santiago M, Valenza MC. Effects of an active intervention based on myofascial release and neurodynamics in patients with chronic neck pain: a randomized controlled trial. Physiother Theory Pract. 2022 Sep;38(9):1145-1152. doi: 10.1080/09593985.2020.1821418. Epub 2020 Sep 15. PMID 32930638